CLINICAL TRIAL: NCT00748488
Title: The ParkFit Study; Effectiveness of an Active Lifestyle Promotion Program for Patients With Parkinson's Disease
Brief Title: Effectiveness of an Active Lifestyle Promotion Program for Patients With Parkinson's Disease
Acronym: ParkFit
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, dr Marten Munneke, PT, Dr, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 50-50310-98-034
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson; Physical Therapy; Physical Activity
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Physical Therapy aimed to promote the level of physical activity
  Interventions: Other: Physical Therapy aimed to improve Physical Activity
- B (Active Comparator): Physical Therapy aimed to move safely
  Interventions: Other: Physical therapy aimed to move safely

INTERVENTIONS:
Other: Physical therapy aimed to move safely — Physical Therapy according to the Dutch guidelines for Physical Therapy in Parkinson's Disease solely focused on safety of movement.
  Duration program: 2 years Maximum number of sessions: 35 per year Duration sessions: 30 minutes
  Arms: B
Other: Physical Therapy aimed to improve Physical Activity — Physical Therapy according to the Dutch guidelines for Physical Therapy in Parkinson's Disease combined with a coaching program aimed to promote the level of physical activity Duration program: 2 years Maximum number of sessions: 35 per year Duration of sessions: 30 minutes
  Arms: A

SUMMARY:
Patients with Parkinson's disease (PD) are heavily inclined towards a sedentary lifestyle. This is caused by a combination of physical impairments and cognitive dysfunction. However, regular physical activity in PD is highly desirable, for two reasons. First, physical activity has positive generic effects in preventing complications such as cardiovascular diseases, type II diabetes mellitus, osteoporosis and certain cases of cancer. Secondly, physical activity has additional disease-specific merits in PD such as depression, sleep disturbances and constipation. These effects lead to raised quality of life. Furthermore, animal studies suggest that physical activity could slow down disease progression.

Simply informing patients about the importance of physical activity is not enough to initiate and maintain an adequate level of physical activity. We propose to develop a physical activity promoting program for sedentary patients with PD in order to raise their level of daily physical activity.

Objective: The first aim of the study is to investigate whether a physical activity promotion program will result in an increase in physical activity in sedentary patients with PD.

The second aim is to demonstrate an increase in physical fitness and quality of life.

DETAILED DESCRIPTION:
no extensive description

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD
* Hoehn and Yahr stage I-III
* Between 40 and 75 years old
* Not meeting the norm for healthy physical activity: the latter being defined according to international standards as either five days a week 30 minutes of moderate-intensity physical activity, or 3 days a week 20 minutes of vigorous-intensity physical activity

Exclusion Criteria:

* Wheel chair bounded
* Severe co-morbidity (e.g. orthopaedic disorders or chronic hart failure)
* Severe cognitive decline, defined as Mini Mental State Examination < 24

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Level of Physical Activity based on the LAPAQ questionnaire | Average of 6, 12, 18 and 24 months

SECONDARY OUTCOMES:
One week diary of physical activity | Average of 6, 12, 18 and 24 months
Level of Physical Activity based on an activity monitor | continuous during 24 months
Physical Fitness (Six Minute Walk Test & Astrand bicycle test) | 12 and 24 months
Quality of Life (PDQ-39) | 6, 12, 18 and 24 months
Mood and Depression (HADS) | 6, 12, 18 and 24 months
Cognition (CANTAB) | 12 and 24 months
disease severity ( Nine Hole Peg test, UPDRS) | 12 and 24 months
Safety(Falls) | monthly
Mobility (Timed up and go test) | 12 and 24 months
Fatigue (FSS) | 6, 12, 18 and 24 months
Medication (questionnaire) | 6, 12, 18 and 24 months
Medical Costs (questionnaire) | 6, 12, 18 and 24 months
Quality of Sleep (SCOPA-sleep) | 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Marten Munneke, Dr., Principal Investigator — UMC st Radboud
Locations (32):
- Netherlands (32):
  - Tergooiziekenhuizen, Hilversum, Postbus 10016
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, Postbus 1101
  - Catharina ziekenhuis, Eindhoven, Postbus 1350
  - Vie Curie Medisch Centrum, Venlo, Postbus 1926
  - Hagaziekhuis, The Hague, Postbus 40551
  - Medisch Centrum Haaglanden, The Hague, Postbus 432
  - Medisch Centrum alkmaar, Alkmaar, Postbus 50
  - Maaslandziekenhuis, Sittard, Postbus 5500
  - Tergooiziekenhuizen, Blaricum, Postbus 900
  - Gelreziekenhuizen, Apeldoorn, Postbus 9014
  - Amphia Ziekenhuis, Breda, Postbus 90157
  - De Gelreziekenhuizen, Zutphen, Postbus 9020
  - Ziekenhuis Gelderse Vallei, Ede, Postbus 9025
  - Elkerliek ziekenhuis, Helmond, Postbus 98
  - Reinier de Graaf Groep, Delft
  - Deventer Ziekenhuis, Deventer
  - Slingeland Ziekenhuis, Doetinchem
  - St. Anna Ziekenhuis, Geldrop
  - Groene Hart Ziekenhuis, Gouda
  - Kennemer Gasthuis, Haarlem
  - Atrium Medisch Centrum, Heerlen
  - Westfriesgasthuis, Hoorn
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Ziekenhuis Bernhoven, Oss
  - Laurentius Ziekenhuis, Roermond
  - Franciscus Ziekenhuis, Roosendaal
  - Erasmus Medisch Centrum, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Sint Franciscus Gasthuis, Rotterdam
  - Vlietland Ziekenhuis, Schiedam
  - Orbis Medisch Centrum, Sittard
  - 't Lange Land Ziekenhuis, Zoetermeer

REFERENCES:
- [Derived] van Nimwegen M, Speelman AD, Overeem S, van de Warrenburg BP, Smulders K, Dontje ML, Borm GF, Backx FJ, Bloem BR, Munneke M; ParkFit Study Group. Promotion of physical activity and fitness in sedentary patients with Parkinson's disease: randomised controlled trial. BMJ. 2013 Mar 1;346:f576. doi: 10.1136/bmj.f576. PMID 23457213
- [Derived] van Nimwegen M, Speelman AD, Smulders K, Overeem S, Borm GF, Backx FJ, Bloem BR, Munneke M; ParkFit Study Group. Design and baseline characteristics of the ParkFit study, a randomized controlled trial evaluating the effectiveness of a multifaceted behavioral program to increase physical activity in Parkinson patients. BMC Neurol. 2010 Aug 19;10:70. doi: 10.1186/1471-2377-10-70. PMID 20723221